CLINICAL TRIAL: NCT04044573
Title: Efficacy of Ultrasound Guided Percutaneous Transperineal Laser Ablation in Benign Prostatic Hypertrophy Patients: Non-Pharmacological Interventional Study
Brief Title: Focal Laser Ablation for Benign Prostatic Hyperplasia
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: University of Rome Tor Vergata (Other)
Responsible Party: Principal Investigator, Guglielmo Manenti, Principal Investigator, University of Rome Tor Vergata
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: R.S.71.18
Record Dates: First submitted 2019-07-11; First posted 2019-08-05 (Actual); Last update posted 2019-08-05 (Actual); Status verified 2019-08

CONDITIONS: Benign Prostatic Hyperplasia; Lower Urinary Tract Symptoms
Keywords: BPH; mpMRI; interventional radiology
MeSH Terms: conditions — Prostatic Hyperplasia; Lower Urinary Tract Symptoms

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

ARMS (1):
- ECHOLASER X4 Socratelite (Experimental): Optic fiber of 300um will be inserted at a distance of 8-10mm from the urethra. Each ablation lasts 6 minutes. Each fiber ablates at an energy of 1800J with a power of 2-3W. Treatment lasts for about 30 minutes.
  Interventions: Procedure: Transperineal Focal Laser Ablation (TPLA)

INTERVENTIONS:
Procedure: Transperineal Focal Laser Ablation (TPLA) — The intervention will take place in an ambulatory setting of the interventional radiology department using the combined Echolaser XVG system. The treatment consists of a local anesthesia to the perineal region. Within each needle, an optic fiber of 300um will be inserted. Each ablation lasts 6 minutes and each fiber ablates1800J at a power of 2-3W. At the end of the ablation there is a pull-back of about 1cm from the original ablation location. According to the dimension of the middle lobe of the prostate, multiple pullbacks can be used. The total ablation is 3600J for 2 fibers (1800J/ fiber) at the power of 2-3W for a total duration of about 30minutes. At the end of the treatment, a 20mg bolus of i.v. corticosteroid is given for anti-edema and anti-inflammatory effects. Antibiotic therapy (Ciprofloxacin 500mg and gastroprotective therapy is given for 5 days. After an adequate amount of time for observation, the patient is dismissed.
  Other Names: Focal Laser Ablation

SUMMARY:
Efficacy of Ultrasound Guided Percutaneous Transperineal Laser Ablation in Benign Prostatic Hypertrophy Patients: Non-Pharmacological Interventional Study

DETAILED DESCRIPTION:
Efficacy of Ultrasound Guided Percutaneous Transperineal Laser Ablation in Benign Prostatic Hypertrophy Patients: Non-Pharmacological Interventional Study

The aim of this pilot study is to evaluate the efficacy of TPLA under US-guidance and the safety and the reproducibility in acute and follow-up.

Objective of the study: Evaluate the efficacy of percutaneous ablative treatment with neodymium laser; the complete profile of safety and tolerability in acute and in the follow-up in patients with Benign Prostatic Hypertrophy by using multiparametric prostate MRI that allows us to evaluate the prostate acutely after treatment and in follow-up. All of the imaging data is correlated with clinical and laboratory data.

Design of the study: Non-pharmacological interventional study. The clinical evaluation will be carried out at three different times:

Time 1: eligibility assessment, signing of informed consent Time 2: admission, laser ablation and control with multiparametric MRI of the post-procedural prostate (T0).

Time 3 Follow up at 3 (T1) -6 (T2) -12 (T3) months from the procedure.

There are various inclusion and exclusion criteria. The inclusion criteria are: over 65 years old, benign prostate hypertrophy (BPH) confirmed by pre-interventional multi-parametric (mpMRI), moderate-elevated surgical risk, presence of urinary obstructive symptoms, signed consent form. Exclusion criteria are: presence of prostate tumor diagnosed by MRI and confirmed by biopsy, urethral stenosis, severe coagulation pathology, ischemic pathology, pacemaker presence, inflammatory pathology in acute phase, presence of 3rd dominant lobe and contraindication to MRI.

Pre-treatment blood chemistry tests:

* Total and fractionated PSA
* Complete blood count with platelet count and leukocyte formula
* Blood coagulation tests
* Urine test - urine culture
* Azotemia
* Creatinine

Technique of performing a percutaneous laser ablation treatment:

The treatments are performed by the radiology team, in an outpatient setting using the Echolaser XVG combined system.

The procedure is performed with the patient in gynecological position, and in safe conditions according to the current legislation for laser treatments (such as protective glasses).

Treatment includes local anesthesia of the perineal region, under ultrasound guidance. At the discretion of the medical team, sedation can be carried out with anesthetic assistance.

2 or 4 needles of 21G, 1 or 2 will be inserted. In each needle a 300 micron optical fiber will be inserted - Elesta s.r.l. - 50041, Calenzano (FI) - Italy, at a distance of 8-10 mm from the urethra. For each ablation, for about 6 minutes, an energy of 1200 J per fiber will be delivered, at the power of 2-5 Watts. At the end the needle and the fiber is retracted for about 1 cm ("pull-back"). Further ablation follows, with delivery and duration and power equal to the previous one. Depending on the size of the middle lobe one or more pull-backs can be made. In total the treatment consists in dispensing up to 1800 J, at the power of 2-5 W for a total duration of 30 minutes.

The laser causes hyperthermia, denaturation and coagulative necrosis of proteins.

The maximum volume treated in a session and the extent of the ablation vary according to the prostatic volume, anatomy and receptivity of the tissue.

At the end of the treatment 20 mg of corticosteroids ev (if not specifically contraindicated by the patient) is administered, for anti-edema and anti-inflammatory purposes. An antibiotic, pain relief and gastroprotective therapy is established for 1 week. After an adequate observation period, the patient will be discharged.

Follow up: The clinical evaluation is carried out at different times

Post procedural follow up:

Immediately after the procedure, a multiparametric prostate MRI is performed, followed by discharge with steroid therapy (prednisone), if not contraindicated, to be scaled and for programming the subsequent follow-up phases.

Post-discharge follow-up:

Specialist examination, suprapubic ultrasound of the urinary tract (with evaluation of the post-residual volume) and multiparametric prostate MRI at 3 months, 6 months and 12 months and subsequent checks according to clinical judgment.

A urine test and any urine culture are attached to each clinical-ultrasound evaluation. At each revaluation the IPSS form and the data collection form is filled out.

ELIGIBILITY:
Inclusion Criteria:

* Over 50 years old
* BPH confirmed by mpMRI
* Uroflowmetry indicating obstructive pathology
* Surgical risk moderate-elevated
* Symptomatology of obstructive pathology (voiding hesitation, intermittent mitt, urinary flow reduction, incomplete emptying of the bladder, post-urination incontinence and irritative symptoms such as urinary frequency, dysuria, nocturia - quantified with IPSS)
* Signature of the information sheet and of the informed consent to the treatment, at the execution of the multiparametric MRI and the administration of the paramagnetic contrast medium.

Exclusion Criteria:

* MRI signs of malignancy confirmed by biopsy investigation
* Urethral stenosis
* Serious coagulation disorders
* Inadequate compliance
* Ischemic pathology in the previous six months
* Presence of pacemakers
* Active phase inflammatory pathology
* Presence of III dominant prostate lobe
* Contraindications to the execution of MRI (claustrophobia, auricular implants, metal prostheses and other contraindications included in the specific informed consent)
* Paramagnetic contrast medium allergy.
* Acute and / or chronic renal failure (GFR <50 mL / min and serum creatinine> 1.5 mg / d)
* Not adequate understanding of the information sheet

Ages: 51 Years to 85 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2018-05-05 (Actual); Primary Completion 2023-04-05 (Estimated); Study Completion 2023-04-05 (Estimated)

PRIMARY OUTCOMES:
Clinical symptoms at 1-yr follow-up evaluated with usual objective and subjective parameters | 12 months
  Improvement of obstructive symptomatology correlated to BPH. The evaluation will be based on urodynamic studies of Qmax, post void and residual volume.
Rate of complication needing re-hospitalisation or reintervention | procedure date to 12 months
  Evaluation of complications post TPLA treatment by MRI.

SECONDARY OUTCOMES:
Reproducibility of Multi-parametric MRI | 12 months.
  Evaluation of multi-parametric MRI of the prostate to quantify and/or preview coagulative necrosis after treatment and evaluate the response to transperineal laser ablation treatment for lower urinary tract symptoms.
Total and post-operative costs during follow-up compared to transurethral resection of the prostate | 12 months
  Calculation and stratification of prodecural costs in in comparison to transurethral resection of the prostate (TURP).
Evaluation of Quality of Life by International Prostate Symptom Score | 12 months
  Evaluation of quality of life quantified by the questionnaire (IPSS)
Evaluation of Quality of Life by International Index of Erectile Function | 12 months
  Evaluation of Quality of Life by International Index of Erectile Function (IIEF)

CONTACTS AND LOCATIONS:
Locations (1):
- Policlinico Tor Vergata (PTV) Foundation: UOC Department of Diagnostic Imaging and Interventional Radiology, Rome, RM, Italy

IPD SHARING:
Plan to Share IPD: Yes
Create an international registry to assess long-term effectiveness of transperineal laser ablation for lower urinary tract symptoms, to assess functional outcomes, to assess safety, to determine baseline patient characteristics, to collect information on possible differences between centres applying treatment of transperineal laser ablation and to explore the optimal treatment indications and possible limitations. It an international prospective observational registry in which data is recorded of patients who are treated with transperineal laser ablation for lower urinary tract symptoms.
Supporting Information: Study Protocol, ICF
Time Frame: This registry will be open for inclusion for five years. Since individual patients will have a follow-up of five years, the total study duration will be 10 years.
Access Criteria: Every accredited centre that performs TPLA procedures, wants to participate and signs the regulatory document and obtains ethical committee approval can participate
URL: http://www.ts-innovations.com/

REFERENCES:
- [Background] Patelli G, Ranieri A, Paganelli A, Mauri G, Pacella CM. Transperineal Laser Ablation for Percutaneous Treatment of Benign Prostatic Hyperplasia: A Feasibility Study. Cardiovasc Intervent Radiol. 2017 Sep;40(9):1440-1446. doi: 10.1007/s00270-017-1662-9. Epub 2017 May 4. PMID 28474112
- [Background] Raz O, Haider MA, Davidson SR, Lindner U, Hlasny E, Weersink R, Gertner MR, Kucharczyk W, McCluskey SA, Trachtenberg J. Real-time magnetic resonance imaging-guided focal laser therapy in patients with low-risk prostate cancer. Eur Urol. 2010 Jul;58(1):173-7. doi: 10.1016/j.eururo.2010.03.006. Epub 2010 Mar 12. PMID 20334965
- [Background] Lindner U, Weersink RA, Haider MA, Gertner MR, Davidson SR, Atri M, Wilson BC, Fenster A, Trachtenberg J. Image guided photothermal focal therapy for localized prostate cancer: phase I trial. J Urol. 2009 Oct;182(4):1371-7. doi: 10.1016/j.juro.2009.06.035. Epub 2009 Aug 14. PMID 19683262
- [Background] Goldberg SN, Grassi CJ, Cardella JF, Charboneau JW, Dodd GD 3rd, Dupuy DE, Gervais D, Gillams AR, Kane RA, Lee FT Jr, Livraghi T, McGahan J, Phillips DA, Rhim H, Silverman SG; Society of Interventional Radiology Technology Assessment Committee. Image-guided tumor ablation: standardization of terminology and reporting criteria. J Vasc Interv Radiol. 2005 Jun;16(6):765-78. doi: 10.1097/01.RVI.0000170858.46668.65. PMID 15947040
- [Background] Bremer C, Kreft G, Roggan A, Filler T, Reimer P. Ex vivo evaluation of novel miniaturized laser-induced interstitial thermotherapy applicators for effective small-volume tissue ablation. Invest Radiol. 2001 Jun;36(6):327-34. doi: 10.1097/00004424-200106000-00005. PMID 11410753
- [Background] Costello AJ, Bowsher WG, Bolton DM, Braslis KG, Burt J. Laser ablation of the prostate in patients with benign prostatic hypertrophy. Br J Urol. 1992 Jun;69(6):603-8. doi: 10.1111/j.1464-410x.1992.tb15631.x. PMID 1379101
- [Derived] Manenti G, Perretta T, Calcagni A, Ferrari D, Ryan CP, Fraioli F, Meucci R, Malizia A, Iacovelli V, Agro EF, Floris R. 3-T MRI and clinical validation of ultrasound-guided transperineal laser ablation of benign prostatic hyperplasia. Eur Radiol Exp. 2021 Sep 17;5(1):41. doi: 10.1186/s41747-021-00239-9. PMID 34532768

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2018-04-23): https://cdn.clinicaltrials.gov/large-docs/73/NCT04044573/Prot_SAP_000.pdf
  • Informed Consent Form (2018-04-23): https://cdn.clinicaltrials.gov/large-docs/73/NCT04044573/ICF_001.pdf